CLINICAL TRIAL: NCT03890159
Title: Effects of Computer Assisted Cognitive Rehabilitation on Patients With Stroke in Attention, Functional Independence and Quality of Life
Brief Title: Effects of Computer Assisted Cognitive Rehabilitation on Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hale Karapolat, Professor in Physical Medicine and Rehabilitation Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Stroke-CACR
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computer Assisted Cognitive Rehabilitation (Experimental): Patients will receive their therapies 1 day a day, 2-3 days a week. The computer-aided cognitive rehabilitation group will perform simulation-based exercises, including exercises related to attention, in a special computer program (Cogniplus TR version) during therapy hours, and patients will progress to the difficulty level automatically. Their performance during this process (response time etc.) will be recorded.
  Interventions: Behavioral: Computer Assited Cognitive rehabilitation
- Conventional Cognitive Rehabilitation (Experimental): The home (paper pen) exercise group will take the necessary exercises on paper suitable for their respective levels and the daily tasks suitable for their functional needs and interests.
  Interventions: Behavioral: Conventional Cognitive Rehabilitation
- Waiting list controls (No Intervention): These patients will get no intervention as means of cognitive rehabilitation, but will get their usual treatments.

INTERVENTIONS:
Behavioral: Computer Assited Cognitive rehabilitation — Patients will receive their therapies 1 day a day, 2-3 days a week. The computer-aided cognitive rehabilitation group will perform simulation-based exercises, including exercises related to attention, in a special computer program (Cogniplus TR version) during therapy hours. The total duration of intervention will be 1 month.
  Arms: Computer Assisted Cognitive Rehabilitation
Behavioral: Conventional Cognitive Rehabilitation — Patients will receive their therapies 1 day a day, 2-3 days a week. The home (paper pen) exercise group will take the necessary exercises on paper suitable for their respective levels and the daily tasks suitable for their functional needs and interests. The total duration of intervention will be 1 month.
  Arms: Conventional Cognitive Rehabilitation

SUMMARY:
This study aims to investigate the effects of computer assisted cognitive rehabilitation and conventional cognitive rehabilitation methods on patients' attention, quality of life and functional independence. Recruiting from 15 patients from each group, patients will be followed up for a month and the outcome measures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with stroke

Exclusion Criteria:

* Problems with sight
* Comorbid neurological disease
* Cognitive impairment prior to stroke
* Neglect Syndrome
* Wernicke or Global aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Stroop test | 1 month
  Stroop test is a quick measurement for ability of color perception and focusing attention Participants are asked to read 112 words with color within 2 min. Then, they are required to tell the color of these 112 words as color-word association. Finally, time of accomplishing task and number of correct read, corrections and errors are examined.
Trail making | 1 month
  Trail making test is used to evaluate the attention and velocity. Participants are asked to sequentially connect 25 circles with number which was written in only one style (Line A), or to sequentially connect 25 circles with number which was written in two styles (Line B). The time used to complete the line A or B and the number of errors and fouls are recorded and analyzed.

SECONDARY OUTCOMES:
Beck Depression Index | Baseline, Month 1
  It is a test frequently used to assess depressive symptoms in chronic diseases. It is comprised of 21 items, 8 of which investigate the somatic symptoms of depression (such as loss of appetite and difficulty sleeping) and 13 of which address the cognitive-affective symptoms of depression (e.g., despair, social withdrawal). The BDI is scored as follows: 0-9: no symptoms; 10-16: mild depression; 17-29: moderate depression; and 30-63: severe depression
Quality of Life Assessment | 1 month
  Medical Outcomes Study 36-item Short Form Survey (SF-36). This is one of the most widely used scales evaluating quality of life. The SF-36 explores eight dimensions of the quality of life "physical function", "physical role", "bodily pain", "general health", "vitality", "social function", "emotional role" and "mental health". All scales were linearly transformed to a 0 to 100 scoring, with 100 indicating most favorable health state and 0 indicating the least favorable health state
Functional Independence | 1 month
  The FIM is a generic and global activity scale that measures an individual's independence in conducting his or her daily fundamental physical and cognitive activities. The FIM measures 81 items in two areas:
  1) physical/motor function (13 items) and 2) cognitive/ psychosocial function (5 items). The items are divided into six subgroups according to activities, four physical and two cognitive. Each item is scored on a scale of one to seven, with "level 1" indicating that the patient needs complete help and "level 7" indicating complete independence. The total FIM score varies between 18 and 126.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186